CLINICAL TRIAL: NCT01314677
Title: Open Label Randomized Trial of Early Assessment of Therapy Response Using 18FDG-PET/CT in Patients With Marginally Resectable Stage IIIA (N2) Non-Small Cell Lung Cancer (NSCLC) Treated With Induction Concurrent Chemoradiation Followed by Resection and Adjuvant Chemotherapy
Brief Title: Fludeoxyglucose F 18 PET/CT Scans in Predicting Therapy Response in Patients With Stage IIIA Non-Small Cell Lung Cancer Undergoing Chemoradiation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects have been accrued to this trial. The PI will no longer be at COH and requests a study withdrawal/closure.
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10012; NCI-2011-00337 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Stage IIIA Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Magnetic Resonance Spectroscopy; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (FDG PET/CT between RT fractions 5-6) (Experimental): Patients undergo a baseline FDG PET/CT scan and receive standard radiotherapy (RT) for 28 fractions with concurrent chemotherapy.
  Patients undergo a FDG PET/CT scan between RT fractions 5-6 (before course 2 of chemotherapy).
  Approximately 6 weeks after completion of CRT, patients undergo a FDG PET/CT scan and undergo standard tumor resection.
  Interventions: Procedure: positron emission tomography/computed tomography (PET/CT); Radiation: fludeoxyglucose F 18
- Group B (FDG PET/CT between RT fractions 10-11) (Experimental): Patients undergo a baseline FDG PET/CT scan and receive standard radiotherapy (RT) for 28 fractions with concurrent chemotherapy.
  Patients undergo a FDG PET/CT scan between RT fractions 10-11 (before course 3 of chemotherapy).
  Approximately 6 weeks after completion of CRT, patients undergo a FDG PET/CT scan and undergo standard tumor resection.
  Interventions: Procedure: positron emission tomography/computed tomography (PET/CT); Radiation: fludeoxyglucose F 18
- Group C (FDG PET/CT between RT fractions 15-16) (Experimental): Patients undergo a baseline FDG PET/CT scan and receive standard radiotherapy (RT) for 28 fractions with concurrent chemotherapy.
  Patients undergo a FDG PET/CT scan between RT fractions 15-16 (before course 4 of chemotherapy).
  Approximately 6 weeks after completion of CRT, patients undergo a FDG PET/CT scan and undergo standard tumor resection.
  Interventions: Procedure: positron emission tomography/computed tomography (PET/CT); Radiation: fludeoxyglucose F 18

INTERVENTIONS:
Procedure: positron emission tomography/computed tomography (PET/CT) — Undergo FDG PET/CT
Radiation: fludeoxyglucose F 18 — Undergo FDG PET/CT
  Other Names: 18FDG; FDG

SUMMARY:
This clinical trial studies fludeoxyglucose F 18 (FDG) positron emission tomography (PET)/computed tomography (CT) in predicting chemoradiation therapy (CRT) failure in patients with stage IIIA non-small cell lung cancer (NSCLC). Diagnostic procedures, such as FDG PET/CT, may help predict CRT failure. Comparing diagnostic results during CRT may help doctors predict a patient's response to treatment and help plan the best treatment

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether early response of the research positron emission tomography (PET)-computed tomography(CT) scan measured by change in Standard Uptake Value (SUV)max relative to baseline scan can predict induction chemoradiation therapy (CRT) failures sooner than post-treatment PET-CT scan.

II. To determine the optimal timing for 18FDG PET-CT that best predicts for induction CRT failure.

SECONDARY OBJECTIVES:

I. To correlate early 18 fludeoxyglucose (FDG) PET-CT response metrics with pathologic response, progression-free survival separately for: induction CRT failures vs. non-failures, or overall survival separately for induction CRT failures vs. non-failures.

OUTLINE: Patients are randomized to 1 of 3 groups.

Patients undergo a baseline FDG PET/CT scan and receive standard radiotherapy (RT) for 28 fractions with concurrent chemotherapy.

GROUP A: Patients undergo a FDG PET/CT scan between RT fractions 5-6 (before course 2 of chemotherapy).

GROUP B: Patients undergo a FDG PET/CT scan between RT fractions 10-11 (before course 3 of chemotherapy).

GROUP C: Patients undergo a FDG PET/CT scan between RT fractions 15-16 (before course 4 of chemotherapy).

Approximately 6 weeks after completion of CRT, patients undergo a FDG PET/CT scan and undergo standard tumor resection.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* All patients with marginally resectable IIIA (N2) NSCLC undergoing induction CRT will be eligible for this imaging trial; patients will be screened by the chest tumor board for entry
* Undergoing or plan to undergo induction chemoradiation

Exclusion Criteria:

* Poorly controlled or uncontrolled diabetes mellitus, with blood glucose > 200 mg/dl
* Have allergies or medical contra-indications to FDG or intravenous (IV) contrast
* Medical contra-indications to obtaining CT or PET scans
* Pre-authorization denial of coverage by insurance providers of clinical staging and restaging PET-CT scans

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Induction therapy failure | 6 weeks after completion of chemoradiation therapy (CRT)
  Defined as any evidence by clinically unresectable disease based on tumor board consensus and review of restaging scans demonstrating locoregional progression or distant metastasis, surgically unresectable disease based on surgical exploration, or suboptimal resection disease still requiring pneumonectomy and still having R1 resection.
Early positron emission tomography (PET) response of group A | Baseline and between standard radiotherapy (RT) fractions 5-6
  Measured by the change in Standard Uptake Value (SUV)max from baseline at the research PET scan in 1 of 3 scheduled time point.
Early positron emission tomography (PET) response of group B | Baseline and between standard radiotherapy (RT) fractions 10-11
  Measured by the change in Standard Uptake Value (SUV)max from baseline at the research PET scan in 1 of 3 scheduled time point.
Early positron emission tomography (PET) response of group C | Baseline and between standard radiotherapy (RT) fractions 15-16
  Measured by the change in Standard Uptake Value (SUV)max from baseline at the research PET scan in 1 of 3 scheduled time point.

SECONDARY OUTCOMES:
Pathologic response | 6 weeks after completion of chemoradiation therapy (CRT)
Progression-free survival | Every 3 months for 2 years and every 6 months thereafter
Overall survival | Every 3 months for 2 years and every 6 months thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Khanh Nguyen, Principal Investigator — City of Hope Medical Center